CLINICAL TRIAL: NCT07283367
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HS-20110 Combination Therapies in Patients With Advanced Colorectal Cancer.
Brief Title: A Phase Ib/II Trial of HS-20110 Combination Therapies in Advanced Colorectal Cancer Patients.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-20110-102
Record Dates: First submitted 2025-12-03; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: CRC

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients in this cohort will receive HS-20110+ Bevacizumab+5-FU/leucovorin in Q2W cycles
  Interventions: Drug: Cohort 1: HS-20110+ Bevacizumab+5-FU/leucovorin
- Cohort 2 (Experimental): Patients in this cohort will receive HS-20110+Bevacizumab+Oxaliplatin+5-FU/leucovorin in Q2W cycles
  Interventions: Drug: Cohort 2: HS-20110+Bevacizumab+Oxaliplatin+5-FU/leucovorin
- Cohort 3 (Experimental): Patients in this cohort will receive HS-20110+Bevacizumab+Oxaliplatin+Capecitabine in Q3W cycles.
  Interventions: Drug: Cohort 3: HS-20110+Bevacizumab+Oxaliplatin+Capecitabine

INTERVENTIONS:
Drug: Cohort 1: HS-20110+ Bevacizumab+5-FU/leucovorin — HS-20110 for IV infusion of various dosage in combination with Bevacizumab+5-FU/leucovorin administered in Q2W doseing cycles
  Arms: Cohort 1
Drug: Cohort 2: HS-20110+Bevacizumab+Oxaliplatin+5-FU/leucovorin — HS-20110 for IV infusion of various dosage in combination with Bevacizumab+Oxaliplatin+5-FU/leucovorin administered in Q2W doseing cycles
  Arms: Cohort 2
Drug: Cohort 3: HS-20110+Bevacizumab+Oxaliplatin+Capecitabine — HS-20110 for IV infusion of various dosage in combination with Bevacizumab+Oxaliplatin+Capecitabine administered in Q3W doseing cycles
  Arms: Cohort 3

SUMMARY:
This is a multicenter, open-label Phase Ib/II clinical study evaluating the safety, tolerability, pharmacokinetics (PK), and efficacy of the HS-20110 combination therapies in Patients with Advanced Colorectal Cancer. "Rolling 6" design would be used to conduct dose escalation part of this study. This study consists of phase Ib and phase II. After RP2D was determined in phase Ib, then a phase II study will be conducted to further evaluate the efficacy, safety, tolerability, and PK of the HS-20110 combination therapies in Patients with mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged ≥ 18 years.
* Participants with pathologically confirmed advanced Colorectal Cancer.
* Participants have at least 1 target lesion other than CNS lesions according to RECIST 1.1.
* MSI was tested to be non-MSI-H, and without BRAF V600E mutation.

Exclusion Criteria:

* Participants have received or are receiving the following treatment:

  1. Anti-tumor drugs within 14 days prior to the first dose of study treatment; any other IMPs or macromolecular anti-tumor drugs within 28 days prior to the first dose of study treatment.
  2. Local radiotherapy within 2 weeks prior to the first dose of study treatment; irradiation of more than 30% of bone marrow or extensive radiotherapy within 4 weeks prior to the first dose of study treatment.
  3. Major surgery within 4 weeks prior to the first dose of study treatment.
  4. Participants previously treated with drugs that are moderate to strong inhibitors or moderate to strong inducers of cytochrome P450 (CYP) 3A4, strong inhibitors or strong inducers of CYP2D6, P-glycoprotein (P-gp), breast cancer resistance protein (BCRP) or drugs with a narrow therapeutic range that are sensitive substrates of P-gp or BCRP within 7 days prior to the first dose of the IMP. Participants who need to receive these drugs during the study period should also be excluded.
  5. Current use of drugs known to prolong the QT interval or that may cause torsade de pointes. Participants who need to receive these drugs during the study period should also be excluded.
  6. Live vaccine or live-attenuated vaccine within 28 weeks prior to the first dose.
* Participants who have any Grade ≥ 2 residual toxicity according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) from prior therapies (except alopecia and residual neurotoxicity).
* Inadequate bone marrow reserve or hepatic and renal functions.
* Participants with a history of severe allergy (such as anaphylactic shock), previous severe infusion reactions, or allergy to recombinant human or murine proteins.
* Participants who are allergic to any component of HS-20110 combination therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or maximum applicable dose (MAD) | From day 1 to one month after the last dose in Phase 1b
Recommended phase 2 dose (RP2D) | From day 1 to one month after the last dose in Phase 1b
Objective response rate (ORR) as per RECIST v1.1 | From day 1 to 3 months after the last patient enrolled in Phase 2

SECONDARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to dose modification or permanent discontinuation, and specific laboratory abnormalities | From the first dose until 90 days after the last dose
Objective response rate (ORR) | From first dose until 3 years after last dose
Incidence of anti-HS-20110 antibody (ADA) | From the first dose until 90 days after the last dose
Drug concentrations of the three components of HS-20110 (including antibody-drug conjugates, total antibody, and payload) | From the first dose until 90 days after the last dose
disease control rate (DCR) | From first dose until 3 years after last dose
duration of response (DoR) | From first dose until 3 years after last dose
progression-free survival (PFS) | From first dose until 3 years after last dose
overall survival (OS) | From first dose until 3 years after last dose